CLINICAL TRIAL: NCT06567418
Title: Effect of In-hospital Initiation of PCSK9i on Clinical Outcomes in Chinese ACS Patients: A Database-based Retrospective Analysis
Brief Title: Retrospective Analysis of the Effect of In-hospital Initiation of PCSK9i on Clinical Outcomes in Chinese ACS Patients
Status: Recruiting | Type: Observational
Sponsor: Yun Dai Chen (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Yun Dai Chen, professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: 2023ESR0000153
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — alirocumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intervention group: patients were treated with alirocumab 75mg combined with statin ± ezetimibe
  Interventions: Drug: alirocumab 75mg/2week
- control group: patients were treated with statin ± ezetimibe only
  Interventions: Drug: statin ± ezetimibe

INTERVENTIONS:
Drug: alirocumab 75mg/2week — patients continually prescribed or stopped alirocumab treatment during the follow-up visit, which depend on physician's clinical decision and patient preference
  Groups: intervention group
Drug: statin ± ezetimibe — patients will be censored at initiation of alirocumab during the follow up visit
  Groups: control group

SUMMARY:
The objective of this study is to investigate the effectiveness of in-hospital initiation of alirocumab combined with statin ± ezetimibe on major cardiovascular events (MACE) in Chinese ACS patients. The main question it aims to answer is:

whether early initiation PCKS9i in hospital could reduce recent cardiovascular event risk in Chinese ACS patients in real-world setting.

Data from CCA Database-Chest Pain Center were screened for all ACS patients from 01-Jan 2021 to 31-Dec 2023. Patients diagnosed with STEMI, NSTEMI or UA at admission were identified at the first step. Then, for intervention group, patients who received alirocumab 75mg combined with statin ± ezetimibe during the ACS hospitalization (including the discharge date) will be included; for control group, patients who received statin ± ezetimibe during the ACS hospitalization will be included. All enrolled patients were required to have at least one documented follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Acute Coronary Syndrome (ACS) upon hospital admission.
* Patients aged 18 years or older.
* Patients who received Alirocumab 75 mg in combination with statin therapy ± Ezetimibe as the intervention group, and those treated exclusively with statin therapy ± Ezetimibe as the control group, either during hospitalization or at discharge.
* Patients with at least one follow-up record.

Exclusion Criteria:

* Patients who received Evolocumab treatment at any time.
* Patients who received Inclisiran treatment at any time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from CCA Database-Chest Pain Center were screened for all ACS patients from 01-Jan 2021 to 31-Dec 2023. Patients diagnosed with STEMI, NSTEMI or UA at admission were identified at the first step. Then, for intervention group, patients who received alirocumab 75mg combined with statin ± ezetimibe during the ACS hospitalization (including the discharge date) will be included; for control group, patients who received statin ± ezetimibe during the ACS hospitalization will be included. All enrolled patients were required to have at least one documented follow-up visit. Patients prescribed with evolocumab at any time will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the risk of MACE within 1 year of follow-up | 12 months
  MACE was defined as the composite of non-fatal myocardial infarction, non-fatal ischemic stroke, all-cause mortality, or any coronary revascularization. Coronary revascularization was limited to procedures occurring at least two weeks after the index date, including PCI and CABG

SECONDARY OUTCOMES:
Percentage reduction of LDL-C levels at 1-month follow-up from baseline | 1 month
  Percentage reduction of LDL-C levels at 1-month follow-up from baseline
Proportion of patient who achieved LDL-C goal (<1.4mmol/L) at 1-month follow-up | 1 month
  Proportion of patient who achieved LDL-C goal (<1.4mmol/L) at 1-month follow-up

OTHER OUTCOMES:
Association between ACS pathway optimization participation and MACE within 1 year follow-up | 12 months
  Association between ACS pathway optimization participation and MACE within 1 year follow-up
Association between ACS pathway optimization participation and LDL-C goal attainment rate at 1-month follow-up | 1 month
  Association between ACS pathway optimization participation and LDL-C goal attainment rate at 1-month follow-up
Percentage reduction of LDL-C levels at 3-month, 6-month follow-up from baseline (if have enough follow-up data on lab test) | 3 months, 6 months
  Percentage reduction of LDL-C levels at 3-month, 6-month follow-up from baseline (if have enough follow-up data on lab test)
LDL-C goal attainment rate (<1.4mmol/L) at 3-month, 6-month follow-up (if have enough follow-up data on lab test) | 3 months, 6 months
  LDL-C goal attainment rate (<1.4mmol/L) at 3-month, 6-month follow-up (if have enough follow-up data on lab test)

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China